CLINICAL TRIAL: NCT01682980
Title: Efficacy of Strength and Aerobic Exercise on Patient-reported Outcomes in Patients With Knee Osteoarthritis - A Randomised Controlled Trial.
Brief Title: Efficacy of Exercise on Quality of Life and Physical Function in Patients With Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Britt Elin Øiestad, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/334
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis; Pain
Keywords: Osteoarthritis; Pain; Exercise; Function; Cartilage quality
MeSH Terms: conditions — Osteoarthritis; Pain; Motor Activity | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Strength training (Experimental): The strength group include progressive strength training and neuromuscular exercises. The inclusion will be performed 2-3 times a week for 12 weeks.
  Interventions: Other: Strength training
- Aerobic exercise (Experimental): The aerobic exercise group will cycle on an ergometer bicycle 2-3 times a week for 12 weeks on moderate loading. The loading will be controlled by a heart rate monitor and is defined as 75% of maximal heart rate (calculated with formula for maximal heart rate reserve).
  Interventions: Other: Aerobic exercise
- Control group (No Intervention): The control group will do as usual.

INTERVENTIONS:
Other: Strength training — The strength training will be delivered 2-3 times per week for 12 weeks, 5-8 repetitions maximum in 3 series. The patients must warm up 5 minutes on an ergometer cycle. The following muscle groups will be trained: Quadriceps and hamstrings, hip muscles (abductors and extensors), calf muscles. A home exercise program will be delivered including one leg exercises and balance exercises. Progression will follow a 2+ principle. For instance, when the study participant is able to perform 2 more repetitions, more loads are required.
  Arms: Strength training
Other: Aerobic exercise — The aerobic exercise program include ergometer cycling for at least 45 minutes 2-3 times a week on 75-80% of max heart rate will be required.
  Arms: Aerobic exercise

SUMMARY:
The overall contribution of this study is to increase the knowledge of the efficacy of strength and aerobic exercise on knee related quality of life, knee pain, and physical function in patients with knee osteoarthritis (OA). Knee OA is one of the most important diseases within musculoskeletal conditions affecting a considerable number of people worldwide. This randomized controlled trial will involve one intervention group delivered strength exercises and one group delivered aerobic exercise (ergometer cycling). The two intervention groups will be compared to a control group undergoing usual care. Cost-effectiveness analysis will be performed comparing the three groups. The study is funded from The Research Council of Norway.

DETAILED DESCRIPTION:
The trial aimed to recruit 207 study participants randomly allocated to three arms. The participants had to have symptomatic knee osteoarthritis verified by grade 2-3 using the Kellgren and Lawrence radiographic classification system, and they had to have knee pain most of the days the last month and fulfil 2/3 of the ACR clinical criteria. Participants with other serious comorbidities or self-reported BMI >35 were included.

The interventions consisted of structured strength training program over 12-14 weeks, and a structured stationary cycling program for 12-14 weeks.

Primary outcome was the KOOS knee-related quality of life subscale at the 1 year follow-up. Secondary outcomes were other patient reported outcomes, muscle strength, and peak oxygen consumption at the 4-month and 1 year follow-up, and over time (1-year).

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 35-70 years
* Clinical knee OA according to the American College of Rheumatology Clinical Criteria
* Kellgren and Lawrence radiographic OA grade 2 and 3 (mild to moderate radiographic OA)

Exclusion Criteria:

* Severe knee OA according to the Kellgren and Lawrence classification (grade 4)
* Other known major musculoskeletal impairments in the lower extremities or the back or prostheses in any joint of the lower extremities
* Known coronary heart diseases or cancer
* Body mass index > 35
* Scheduled for surgery in any joint
* Known mental or psychologic diseases
* Known drug abuse
* Persons who already perform sports related moderate physical activity more than two times a week
* Contraindications for magnetic resonance imaging (specific point list at Oslo University Hospital, radiographic department)
* Not speaking Norwegian language

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2013-03; Primary Completion 2023-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Knee-related quality of life | 1 year
  Primary outcome for the study will be the quality of life subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) (0-100 scale). 0 is very poor knee-related quality of life, while 100 indicates normal knee-related quality of life.

SECONDARY OUTCOMES:
Knee function | 4 months and 1 year
  The KOOS is a self-administered knee-specific questionnaire containing 5-item Likert scales on pain, other symptoms, activities of daily living (ADL), function in sports and recreation and knee-related quality of life (QOL). Each scale goes from 0-100, 0 indicating worse function and 100 representing normal function.
Health-related quality of life | 4 months and 1 year
  Euro Quality of life 5 dimensions 5 level (EQ-5D-5L) will be used to measure health related quality of life. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EuroQol (EQ) Visual analogue scale (VAS) records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
Radiographic osteoarthritis progression | 2 years
  Conventional x-rays will be used to assess radiographic progression of osteoarthritis

OTHER OUTCOMES:
Isokinetic muscle strength | 4 months and 1 year
  Isokinetic muscle strength will be measured in a Biodex6000 machine. The participants sit in a standardised position and flex/extend their knees at 60 degrees/second. The peak torque value of the five repetitions is recorded.
Maximal oxygen consumption (VO2max) | 4 months and 1 year
  VO2max is measured using an incremental ramp test procedure on a stationary bike, designed to achieve supramaximal workloads within ~4-6 min. The workload was increased by 25 watts every 30 second to total exhaustion.
Self-efficacy for pain | 4 months and 1 year
  Arthritis self-efficacy scale (ASES) was included to measure self-efficacy for pain. A modified version of ASES containing 11 questions regarding the patient's certainty to perform various tasks related to pain and symptoms, where each item is rated from 1 (very uncertain) to 5 (very certain) was used.
Total knee replacement | 5 years
  We will register continuously numbers of total knee replacements during the follow-up years.

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Killingmo RM, Oiestad BE, Risberg MA, Maas E, Grotle M. Cost-effectiveness of strength exercise or aerobic exercise compared with usual care for patients with knee osteoarthritis: secondary results from a multiarm randomised controlled trial in Norway. BMJ Open. 2024 May 23;14(5):e079704. doi: 10.1136/bmjopen-2023-079704. PMID 38803266
- [Derived] Oiestad BE, Aroen A, Rotterud JH, Osteras N, Jarstad E, Grotle M, Risberg MA. The efficacy of strength or aerobic exercise on quality of life and knee function in patients with knee osteoarthritis. A multi-arm randomized controlled trial with 1-year follow-up. BMC Musculoskelet Disord. 2023 Sep 8;24(1):714. doi: 10.1186/s12891-023-06831-x. PMID 37684597
- [Derived] Oiestad BE, Osteras N, Frobell R, Grotle M, Brogger H, Risberg MA. Efficacy of strength and aerobic exercise on patient-reported outcomes and structural changes in patients with knee osteoarthritis: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2013 Sep 12;14:266. doi: 10.1186/1471-2474-14-266. PMID 24028201

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT01682980/SAP_001.pdf